CLINICAL TRIAL: NCT02792868
Title: Biological Phosphocalcic Metabolism and Coronary Artery Calcifications
Acronym: BIOCAC
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 2015.02
Record Dates: First submitted 2016-05-26; First posted 2016-06-08 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood 24h urines
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patient: patient with cardiovascular risk (moderate)
  Interventions: Other: 24 h urines analyses

INTERVENTIONS:
Other: 24 h urines analyses — patient collects urines during 24h

SUMMARY:
Study a sample of patients in primary prevention, moderate cardiovascular risk (n = 83 patients), with normal, non-diabetic renal function. The investigators quantify the phophocalcic intake and excretion, realizing a food examination and a urine collection of 24 particular. The investigators will measure plasma levels of FGF23 serum calcium, phosphatemia, the investigators will calculate the tubular reabsorption of phosphate. The investigators will conduct a quantitative assessment of coronary calcification by a non-injected CT scan, measuring semi automated way Agatston calcium score. There will be an analysis of collinearity. An adjustment will be made for confounding variables in a generalized linear regression model.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization for a cardiovascular check in the Detection Centre and the Atherosclerosis Prevention (CHU Rangueil Toulouse)
* In primary prevention of coronary heart disease
* Introducing an intermediate cardiovascular risk according to the European SCORE equation, that is to say, a risk of cardiovascular death at 10 years greater than or equal to 1% and less than 5%
* signed the informed consent,

Exclusion Criteria:

* Chronic renal failure patients with an estimated GFR less than 60 mL / min / 1.73m2, due to alterations in phosphate metabolism,
* Patients receiving glucose-lowering therapy,
* Patients with a fasting blood glucose greater capillary or equal to 1.10 g / l, confirmed by a plasma glucose greater than or equal to 1.10g / l.
* The diuretic therapy patients (due to a change in urinary electrolytes)
* HIV-positive patients for HIV, antiretroviral (due to a change in urinary electrolytes)
* Pregnant women,
* Patients under judicial protection, guardianship or trusteeship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with cardiovascular risk
Sampling Method: Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2016-04; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
plasma levels of FGF23 according to the calcium score, determined by an ELISA method | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Jean FERRIERES, Principal Investigator — CHU RANGUEIL
Locations (1):
- Chu Rangueil, Toulouse, France